CLINICAL TRIAL: NCT02239185
Title: Laparoscopic Inguinal Hernia Repair in Infancy and Childhood; a Prospective Controlled Randomized Study of Two Different Technique
Brief Title: Laparoscopic Inguinal Hernia Repair in Infancy and Childhood
Acronym: LIHR-2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Rafik Shalaby, professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-2014; RAFIK-2014 (Registry Identifier: Al Azhar University)
Record Dates: First submitted 2014-02-26; First posted 2014-09-12 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Congenital Inguinal Hernia
Keywords: Laparoscopy; purse string; hernial sac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hernial sac ligation in continuity (Other): laparoscopic closure of hernia sac in continuity using 3 - 0 non-absorbable purse-string suture. Two 3-mm.needle holders are used for intracorporeal insertion of purse string suture around the opened IIR with intracorporeal knot tying.
  Interventions: Procedure: Hernial sac ligation in continuity
- Hernial sac disconnection (Other): circumferential incision on the peritoneum at internal inguinal ring (IIR) with separation of hernia sac from the peritoneum. The proximal part of the sac will be sutured using non-absorbable 3-0 prolene on round body needle.
  Interventions: Procedure: Hernial sac disconnection

INTERVENTIONS:
Procedure: Hernial sac ligation in continuity — Laparoscopic closure of hernia sac at internal inguinal ring in continuity using 3 - 0 non-absorbable purse-string suture. The spermatic vessels and vas deferens are well visualized and protected during the suture. In all cases, hydro dissection can be done by injection of saline to separate the peritoneum from cord structures. Two 3-mm.needle holders are used for intracorporeal insertion of purse string suture around the opened IIR with intracorporeal knot tying. The stitches included the peritoneum and the underlying muscular tissue lateral to the spermatic cord. The procedure is modified in children with a dilated internal ring.
  Other Names: Purse string suture around IIR leaving the sac in continuity
  Arms: Hernial sac ligation in continuity
Procedure: Hernial sac disconnection — Circumferential incision on the peritoneum at IIR will be started to separate hernia sac from the peritoneum. Initial disconnection of the vas and vessels will be done and then the peritoneum posterior to the internal ring will be divided and then the anterior disconnection will be carried out. Saline can be injected to separate the peritoneum from cord structures (hydro dissection). Care is taken not to damage the vas and vessels by handling them. Then the proximal part of the sac will be sutured using non-absorbable 3-0 prolene on round body needle.
  Other Names: Laparoscopic disconnection of the hernial sac at IIR
  Arms: Hernial sac disconnection

SUMMARY:
Aim of the study The aim of this study is to test the hypothesis that during laparoscopic hernia repair, disconnection of the hernial sac along with suture ligation of the neck is better than transperitoneal purse string suture around the hernial sac at the neck leaving the sac in continuity. Also to compare the two different laparoscopic techniques as regards operative time, recurrence rate, hydrocele formation, and other possible complications as bleeding, hematoma, injury of the vas and testicular atrophy and post-operative cosmetic results.

..

DETAILED DESCRIPTION:
Ethical Consideration:

The protocol will be discussed and approved for clinical study by the Ethical Research Committee of our University. The procedures and the aim of the study are clearly explained to the patient and the family. A written informed consent is obtained before enrollment of the patients into the study. The family refusal to give consent for laparoscopic hernia repair by either technique does not deprive the patient from getting surgical care by open herniotomy

• In the 2 groups, after induction of general endotracheal tube anesthesia, the patient is positioned supine in Trendelenburg's position. Insertion of the main umbilical port [5-mm] by open technique will be done for 5-mm 30° telescope, then pneumoperitoneum will be created to a pressure of 8-12 mmHg.

Laparoscopy will be used for initial visualization of the pelvis and internal inguinal rings on both sides. In group I, the laparoscopic hernia repair will be done according to a technique described by Scheir Two 3-mm trocars are inserted under laparoscopic guidance at the level of umbilicus in mid-clavicular line on either side as working ports unilateral hernia, on the side of hernia can be little higher and opposite side little lower, for better triangulation. In infants and small babies, the working ports are placed little higher than the level of umbilicus.

Non absorbable 3-0 Prolene suture is used in all patients after its shortening to 8cm.length.

Group I, laparoscopic closure of hernia sac at internal inguinal ring in continuity using 3 - 0 non-absorbable purse-string suture. The spermatic vessels and vas deferens are well visualized and protected during the suture. In all cases, hydro dissection can be done by injection of saline to separate the peritoneum from cord structures. Two 3-mm.needle holders are used for intracorporeal insertion of purse string suture around the opened IIR with intracorporeal knot tying. The stitches included the peritoneum and the underlying muscular tissue lateral to the spermatic cord. The procedure is modified in children with a dilated internal ring. Ligature of the hernia sac at internal inguinal ring (IIR) is inadequate in such cases. Here, laparoscopic narrowing of IIR by few interrupted sutures will be done.

Group II, circumferential incision on the peritoneum at IIR will be started to separate hernia sac from the peritoneum. Initial disconnection of the vas and vessels will be done and then the peritoneum posterior to the internal ring will be divided and then the anterior disconnection will be carried out. Saline can be injected to separate the peritoneum from cord structures (hydro dissection). Care is taken not to damage the vas and vessels by handling them. Then the proximal part of the sac will be sutured using non-absorbable 3-0 prolene on round body needle. Closure: In both groups, supra-umbilical incision will be closed with polyglycolic acid 3-0 suture. Three mm trocar sites will be approximated with the steri-strips.

ELIGIBILITY:
Inclusion Criteria:

Bilateral congenital inguinal hernia (CIH), recurrent cases, unilateral cases with questionable other side, parental request and cases with CIH associated with umbilical hernia.

Exclusion Criteria:

Hernia of canal of Nuck in females, Inguinal hernia with undescended testis, Parental refusal, Contraindications for laparoscopy as lower major abdominal surgery

Ages: 6 Months to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Recurrence | At 3 and 6 months post operatively
  All Patients will be subjected to post operative clinical examination and scrotal U/S for assessment of the recurrence. Recurrence is identified by visual of a bulg at the site of hernia on crying and the presence of defect more than 4 mm. In diameter

SECONDARY OUTCOMES:
Operative time | intra operative time is measured from skin incision to skin closure
  The operative time will be measured by minutes in both group. The operative time is measured from skin incision to skin closure. It does not enclude induction and recovery of anesthesia.
Post operative hydrocele formation | at 1 and 3 months post operatively
  Post operative hydrocele formation is evaluated by clinical and U/S examination. It is measured by milliter of fluids in the tunica vaginalis around the testis

CONTACTS AND LOCATIONS:
Overall Officials: Rafik MI Shalaby, MD, Principal Investigator — Al-Azhar University
Locations (1):
- Rafik Shalaby, Cairo, Egypt

REFERENCES:
- [Background] Shalaby R, Ibrahem R, Shahin M, Yehya A, Abdalrazek M, Alsayaad I, Shouker MA. Laparoscopic Hernia Repair versus Open Herniotomy in Children: A Controlled Randomized Study. Minim Invasive Surg. 2012;2012:484135. doi: 10.1155/2012/484135. Epub 2012 Dec 27. PMID 23326656